CLINICAL TRIAL: NCT01673542
Title: Evaluating the Effectiveness of Dermal Analgesia Provided by the Application of Lidocaine and Prilocaine Cream 5% on the Puncture Site of Axillary Blocks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EMLAX 2012-001976-13
Record Dates: First submitted 2012-07-09; First posted 2012-08-28 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Surgery Scheduled

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine-Prilocaine 5% (Experimental)
  Interventions: Drug: Lidocaine-Prilocaine 5%
- Dexeryl (Placebo Comparator)
  Interventions: Drug: DEXERYL

INTERVENTIONS:
Drug: Lidocaine-Prilocaine 5%
  Arms: Lidocaine-Prilocaine 5%
Drug: DEXERYL
  Arms: Dexeryl

SUMMARY:
Prospective Study, monocentric, controlled, randomized study. Evaluating the effectiveness of dermal analgesia provided by the application of Lidocaine and Prilocaine Cream 5% on the puncture site of axillary blocks.Our study includes 70 patients. Number of subjects required for a 50% difference with the standard deviation of the control group, a significance level of 5% for a 80% power, it takes 23 people per group. Objective power of 90% obtained with 35 patients per group.

The expected benefit is the reduction of pain at the skin puncture during the realization of BAX.

Improving professional practice and quality care

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalized for upper extremity surgery scheduled
* Having an axillary block anesthesia.
* Free subject, without subordination or guardianship
* Patients undergoing a social security system or benefiting through a third party
* Informed consent and signed by the patient after clear and honest information on the study

Exclusion Criteria:

* Age < 18 years
* Hypersensitivity to lidocaine, prilocaine, to one of the excipients, castor oil and its derivatives
* Hypersensitivity to local anesthetics of the amide
* Congenital Methemoglobinemia
* Porphyrias
* Glucose-6-phosphate dehydrogenase
* Hypersensitivity to any component of Dexeryl ®
* Disorders of atrioventricular conduction requiring permanent pacing not yet realized.
* Epilepsy uncontrolled by treatment
* Patients on anticoagulants
* Skin infection from the puncture site
* Patients with psychiatric disorders or dementia
* Cons-indication for infusion Isofundine ®:
* Severe congestive heart failure
* anuria
* oligoanuria
* Fluid retention
* hyperkalemia
* hypercalcemia
* Metabolic alkalosis
* Patients not receiving a social security system or not qualifying through a third party
* People receiving more protection ie minors, persons deprived of liberty by a judicial or administrative decision, guests staying in a hospital or office, adults under legal protection,
* Pregnant or nursing women, women of childbearing age who do not have effective contraception (hormonal / mechanical: oral, injectable, transdermal, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, oophorectomy total )

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Compare the VAS groups of Lidocaine-Prilocaine 5% and Dexeryl ®
  The main objective of the study is to compare the VAS (visual analogue scale) between groups of Lidocaine-Prilocaine 5% and Dexeryl ® in pain at the skin puncture for producing a block in patients undergoing axillary to an upper extremity surgery

SECONDARY OUTCOMES:
evaluation pain
  - Pain during injection of mepivacaine, measured by a visual analog scale (VAS) from 0 to 100 mm,
satisfaction
  - Assessment of satisfaction of anesthetists
success
  The success rate of the block defined by the absence of recourse to another anesthetic technique for inadequate analgesia (the use of hypnotic anxiolytic

CONTACTS AND LOCATIONS:
Locations (1):
- Service Anesthésie-Réanimation, Poitiers, France